CLINICAL TRIAL: NCT03858439
Title: Dietary Intervention in Patients With ADPKD on Tolvaptan: Urine Output and Quality of Life
Brief Title: Dietary Intervention in ADPKD on Tolvaptan
Acronym: DIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Peter Margetts, Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v1
Record Dates: First submitted 2019-02-04; First posted 2019-02-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Polyuria; Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polyuria; Polycystic Kidney, Autosomal Dominant | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Single group before / after dietary intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Single arm study. All participants will receive dietary intervention.
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary — Low sodium, low protein dietary recommendation

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common inherited renal disorder. Tolvaptan has been approved in Canada as a treatment for ADPKD. Tolvaptan is an arginine vasopressin receptor antagonist which has been shown to decrease the progression of ADPKD. The main side effect of this treatment is increased urine output which leads to cessation of therapy in about 20% of patients. Low solute (low sodium, low protein) diet may alleviate this side effect. This is a single arm before / after study of dietary intervention on urine output and quality of life in ADPKD patients on a stable dose of tolvaptan.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common inherited renal disorder affecting 12.5 million persons worldwide, and impacting approximately 35,000-66,000 Canadians. An estimated 45% to 70% of patients with ADPKD progress to end-stage renal disease by age 65 years.

Tolvaptan has been approved in Canada as a treatment for ADPKD. Tolvaptan was discovered in Japan by Otsuka Pharmaceutical and was first approved there for ADPKD in 2014. The Health Canada approval of Tolvaptan is based on the results of the pivotal Phase 3 randomized, double-blind and placebo-controlled TEMPO 3:4 Trial, the largest study conducted to date in adults with ADPKD.

The treatment of ADPKD had previously been symptomatic with the aim of reducing morbidity and mortality associated with disease manifestations. This changed with the publication of the TEMPO 3:4 trial, which proved the efficacy of the arginine vasopressin (AVP) V2 receptor antagonist tolvaptan in decreasing the progression of CKD. In this trial, 1445 patients with ADPKD eGFR > 60 were randomized to receive either placebo or tolvaptan in a split-dose regimen of 45 mg in the morning and 15 mg in the afternoon, up titrated to 90/30 mg as tolerated. The REPRISE study investigated the value of tolvaptan in 1300 patients with lower levels of eGFR (25-65 mL/min/1.73 m2).

AVP plays a major role in the pathogenesis of cysts in ADPKD via cAMP stimulation. The AVP antagonist blocks V2 receptors in collecting ducts and therefore blocks the concentrating ability of the tubule. This leads to increased urine volume. Recently, it has been demonstrated that this increased urine volume is related to solute excretion. Therefore, it seems possible that dietary modification to decrease solute intake (salt, protein) would decrease the urine volume in patients taking tolvaptan.

The most common side effect of AVP antagonist is increased renal water excretion which presents as polyuria, nocturia, increased thirst, and dry mouth. The daily urine volumes 5 days after starting different split doses of tolvaptan (15/15, 30/0, 30/15, 30/30 mg) in a preliminary phase 2 study were 4 to 6 L. In the treatment of hyponatremia and heart failure (another indication for tolvaptan therapy), a meta-analysis found an average increase in water clearance of only 68 mL/h after tolvaptan treatment. This more modest increase in urine output may be related to the low sodium diet most of these patients should be adhering to.

ELIGIBILITY:
Inclusion Criteria:

1. Patients seen in the Hamilton Nephrology Genetics Clinic with a diagnosis of ADPKD taking tolvaptan
2. Able to provide informed consent
3. On maximal tolerated dose of tolvaptan for at least 3 months

Exclusion Criteria:

1. Serum sodium > 135 mmol/L
2. Patients with evidence of non-compliance (not completing monthly blood work required while on tolvaptan therapy).
3. Unlikely to continue in Hamilton Nephrology Genetics Clinic for at least 6 months (planned dialysis initiation, transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urine volume | Change from baseline to 3 months
  24-hour urine volume in ml.

SECONDARY OUTCOMES:
Change in ADPKD-IS | Change from baseline to 3 months
  Autosomal dominant polycystic kidney disease impact score - quality of life. Eighteen items, score from 18 to 90 with higher values reflecting lower quality of life
Change in Nagasaki Diabetes Insipidus Questionnaire | Change from baseline to 3 months
  Validated measure of polyuria on quality of life. Subset of questions 1-10 will be used (Questions 11-12 relate to therapy with DDAVP). Score from 10 to 40 with higher scores reflecting worse quality of life.
Change in urine total solute | Change from baseline to 3 months
  Urine total solute measured by (urine sodium + urine urea) * urine volume

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No